CLINICAL TRIAL: NCT05134766
Title: Retrospective Evaluation of Clinical, Virological and Serological Data in Patients With Mild Acute Upper Respiratory Tract Infections
Status: Completed | Type: Observational
Sponsor: Complex Medical Centre Deli Klinika (Other)
Collaborators: Herb-Pharma Sk, s.r.o. (Unknown); Medix Clinical & Academic Research Consulting (Unknown)
Responsible Party: Sponsor
Other Study IDs: CMA-R2107
Record Dates: First submitted 2021-11-15; First posted 2021-11-26 (Actual); Last update posted 2021-11-26 (Actual); Status verified 2021-11

CONDITIONS: Acute Upper Respiratory Tract Infection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- PCR positive: Those with a condition of the first SARS-CoV-2 PCR test result was positive. Based on data recorded in the period between 01 January 2021 to 30 June 2021
  Interventions: Other: Observation only
- PCR negative: Those with a condition of the first SARS-CoV-2 PCR test result was negative. Based on data recorded in the period between 01 January 2021 to 30 June 2021
  Interventions: Other: Observation only
- IgA/IgG positive: Those with a condition of the first IgA or IgG test result was at least once positive.
  Interventions: Other: Observation only
- IgA/IgG negative: Those with a condition of the first IgA and IgG test results were both negative
  Interventions: Other: Observation only
- Prevention only: Those with a condition of the first SARS-CoV-2 PCR test result was negative AND IgG /IGA negative.
  Interventions: Other: Observation only
- W/Symptoms: Those that reported at least one positive symptom. Based on data recorded in the period between 01 January 2021 to 30 June 2021
  Interventions: Other: Observation only

INTERVENTIONS:
Other: Observation only — Based on type of SOC applied and the type of CAM products by subject's own decison

SUMMARY:
Retrospective analysis with subgroup evaluation

Primary objectives of the data analysis study:

1 Retrospective analysis of the symptoms and quality of life data of patients with mild, acute (<96 hours) upper respiratory symptoms based on the results of standard health assessment questionnaires used at the institution, over a period of 10-15 days after the SARS CoV-2 PCR test.

Secondary objectives

1 Retrospective assessment of the upper respiratory tract symptoms and quality of life and serological parameters of the contact persons with confirmed close exposure to SARS CoV-2 PCR positive patients (based on the results of the standard health assessment questionnaires used at the institution in the period of 10-15 days after the SARS CoV-2 PCR test)

The retrospective analysis also includes an assessment of the pharmacological and supplementary therapies used in patients presenting with mild, acute (<96 hours) upper respiratory symptoms and SARS CoV-2 positive contacts, as well as the incidence of SARS CoV-2 virus infection in contacts confirmed by PCR test (based on values measured within 48 hours and 10-15 days later), and an analysis of patients' serological data.

DETAILED DESCRIPTION:
1. Symptoms and quality of life data of patients with mild, acute upper respiratory symptoms in the stated period, as recorded in standard health assessment questionnaires used at the institution. Symptoms and quality of life parameters recorded during the course of acute mild upper respiratory disease based on the health assessment questionnaires used at the institution and international standard upper respiratory questionnaires (revised " CMC Déli Klinika - Clinical Data, Health and Risk Assessment Related to the SARS CoV-2 Tests" questionnaire and the WHO-protocol_2019-nCoV-Seroepidemiology-2020.1 and WURSS based on "Wisconsin Upper Respiratory Symptom Survey - WURSS-24 - Daily Symptom Report".
2. Clinical laboratory data: Results of the SARS CoV-2 PCR and serological tests over a 15-day period. As an additional cohort, contact persons with close exposure, who were asymptomatic or presenting with mild upper respiratory symptoms, in whose case the SARS CoV-2 virus was detected by PCR within 48 hours and the proximity of SARS CoV-2 PCR positive patients can be considered as potential exposure.

The study was conducted between 01 January 2021 to 30 June 2021, using data from patients presenting at the CMC Déli Klinika. Data analysis for research purposes includes a critical analysis of the results of the enrollment tests, the so-called (baseline data) laboratory data and the results from the online (follow-up) symptom diaries.

For all persons presenting at the institution, it should be confirmed during the standard consent procedure of the clinic that the CMC Déli Klinika conducting the data collection will treat patient documents and data in strict confidence. In addition, all personal data, especially sensitive data related to the health of the research participants, must be handled in accordance with GDPR 2016/679 and all related local requirements.

The data collection perod is 1 January 2021 to 30 June 2021, using data from patients presenting at the CMC Déli Klinika. Data analysis for research purposes includes a critical analysis of the results of the enrollment tests, the so-called (baseline data) laboratory data and the results from the online (follow-up) symptom diaries.

Due to the retrospective observational nature of the study, the analysis will be descriptive/exploratory. Available data from all patients who meet the inclusion criteria will be included in the analysis. The subgroups will be analyzed in an exploratory way (e.g. by age, gender, medications used and other supplementary therapies, and by relevant subgroups). The analysis plan is to be developed at an analytical statistical meeting after the primary analysis of the data for the period under review. One of the variables in the study is the change in the revised WURSS-24 scale score on days 10-15 compared to the baseline 2-day value, and its change in the 2-10 day period under review. The change will be analyzed by descriptive statistical methods, there will be no formal hypothesis testing. The results of the statistical tests performed will be interpreted descriptively. Continuous data will be described by statistical estimates (mean, standard deviation, minimum and maximum, mode, median). Categorical data will be characterized by absolute frequency and percentage. The parameters related to the research study objectives will be described descriptively, and the time course and characteristic extreme values of each data set will be presented. According to the applied treatment, the data will be compared by t-test in the case of two groups and by ANOVA in the case of more than 2 groups. The change over time will also be presented graphically. For the proportion of PCR-positive patients confirmed by standard diagnostic procedure, the proportion of COVID-positive patients confirmed by PCR and PCR-positive contact persons on days 10-15 and the related 95% confidence interval will be determined. The ratios measured in each treatment subgroup will be compared by Chi-square test.

For quality of life questions used by the institution, the quality of life will be evaluated on a QoL scale. The results of the questionnaires will be summarized separately for each subgroup by time, using descriptive statistics. For continuous variables, the number of cases, mean, standard deviation, median, minimum and maximum values will be presented. For categorical variables, the case number and frequency will be presented.

In the course of its healthcare services, the institution provides medical and health data related to patients in accordance with the data protection standards, confidentiality and local/regional/national requirements. All records and patient documents being kept confidential. During the retrospective analysis, the data will be stored exclusively in a coded form according to the institution's database, anonymously. In order to process the data, they will be entered and checked by qualified staff in accordance with the daily standard routine. The inspection of the clinical data of the retrospective survey will be performed for the purpose of verification by a designated independent clinical research specialist at the study site. The statistical evaluation of the data and the comparison of the results of each subgroup will be carried out with the involvement and under the guidance of a specialist statistician. Descriptive statistical methods, as well as the formation of relevant subgroups for each parameter and the drug and supplementary therapies used to treat symptoms, and comparative analysis of cohort data. Data will be analyzed anonymously, aggregated and by subgroups.

The institution conducting the research is responsible for submitting an application, in an appropriate method and form, for the ethical authorization of the retrospective analytical research. In accordance with the relevant rules of procedure, a copy of the submitted documentation as well as the source data used and its database will be archived by the principal investigator.

ELIGIBILITY:
Inclusion Criteria:

* Groups of patients who volunteer at the institution to have laboratory testing or laboratory sampling who

  * present with symptoms of mild respiratory infection and have these symptoms for no more than 96 hours
  * are at least 18 years old
  * have requested and have had standard laboratory tests, blood sampling or SARS-CoV sampling provided by the institution in accordance with the institution's procedures,
  * entered evaluable responses at least three times on the standard online health questionnaires provided by the institution,
  * participated in at least 2 SARS CoV-2 sampling tests,
  * and for whom no such clinical condition or other reason was identified during the data review and assessment by the principal investigator that could affect the integrity of the data

Exclusion Criteria:

* Subjects will be excluded from the analysis who:

  * Have symptoms suggestive of moderate to severe condition:

    * breathing rate: > 21/min AND/OR
    * extra oxygen demand (e.g. peripheral oxygen saturation measured on site <96%)
    * AND/OR clinical or radiological signs of pneumonia, or other conditions considered severe by the specialist, clinician or requiring hospitalization
    * or were also hospitalized in connection with the COVID-19 disease
  * Have infection-specific or COVID-19 disease-specific symptoms for more than 96 hours when first presenting, or
  * Have a history of chronic ethyl consumption or smoking >20 cigarettes per day, or suspected COPD

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The objective of the research is retrospective data analysis based on the institution's own data, with their anonymous post-processing and analysis by subgroups, with special regard to the self-reported health assessment data on acute upper respiratory symptoms of the participating patients, their follow-up, and the results of relevant standard laboratory tests performed in the study period in the population determined on the basis of the selection criteria.
Sampling Method: Non-Probability Sample
Enrollment: 380 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Change in conditions and symptoms | baseline and every other day over a period of up to 15 days after the SARS CoV-2 PCR test competed.
  Assessment of change in condition, change in symptoms based on standard completed online symptom diaries, based on retrospective analysis of the symptoms and quality of life data results of standard health assessment questionnaires used at the institution.

SECONDARY OUTCOMES:
Results of repeated PCR and serological tests | baseline (d0-d2) and follow-up 10-15 days later
  serological parameters of the SARS CoV-2 PCR positive patients and negative subjects

OTHER OUTCOMES:
Pharmaco-therapies and supplementary therapies | baseline (d0-d2) and a control 10-15 days later
  Assessment of the composition and charaterictics of pharmacotherapies and supplementary (CAM) therapies used in patients with mild, acute upper respiratory symptoms at baseline and SARS CoV-2 and similar that to contacts, as well as the incidence of SARS CoV-2 virus infection in contacts confirmed by the follow-up PCR test.

CONTACTS AND LOCATIONS:
Overall Officials: Botond Lakatos, MD, Principal Investigator
Locations (1):
- Complex Medical Centre Deli Klinika, Budapest, Hungary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Goc A, Sumera W, Rath M, Niedzwiecki A. Phenolic compounds disrupt spike-mediated receptor-binding and entry of SARS-CoV-2 pseudo-virions. PLoS One. 2021 Jun 17;16(6):e0253489. doi: 10.1371/journal.pone.0253489. eCollection 2021. PMID 34138966
- [Background] Droebner K, Ehrhardt C, Poetter A, Ludwig S, Planz O. CYSTUS052, a polyphenol-rich plant extract, exerts anti-influenza virus activity in mice. Antiviral Res. 2007 Oct;76(1):1-10. doi: 10.1016/j.antiviral.2007.04.001. Epub 2007 May 15. PMID 17573133
- [Background] Di Pierro F, Derosa G, Maffioli P, Bertuccioli A, Togni S, Riva A, Allegrini P, Khan A, Khan S, Khan BA, Altaf N, Zahid M, Ujjan ID, Nigar R, Khushk MI, Phulpoto M, Lail A, Devrajani BR, Ahmed S. Possible Therapeutic Effects of Adjuvant Quercetin Supplementation Against Early-Stage COVID-19 Infection: A Prospective, Randomized, Controlled, and Open-Label Study. Int J Gen Med. 2021 Jun 8;14:2359-2366. doi: 10.2147/IJGM.S318720. eCollection 2021. PMID 34135619
- [Background] El-Anwar MW, Elzayat S, Fouad YA. ENT manifestation in COVID-19 patients. Auris Nasus Larynx. 2020 Aug;47(4):559-564. doi: 10.1016/j.anl.2020.06.003. Epub 2020 Jun 15. PMID 32586739
- [Background] Rosas-Salazar C, Kimura KS, Shilts MH, Strickland BA, Freeman MH, Wessinger BC, Gupta V, Brown HM, Rajagopala SV, Turner JH, Das SR. SARS-CoV-2 infection and viral load are associated with the upper respiratory tract microbiome. J Allergy Clin Immunol. 2021 Apr;147(4):1226-1233.e2. doi: 10.1016/j.jaci.2021.02.001. Epub 2021 Feb 9. PMID 33577896
- [Background] Ra SH, Lim JS, Kim GU, Kim MJ, Jung J, Kim SH. Upper respiratory viral load in asymptomatic individuals and mildly symptomatic patients with SARS-CoV-2 infection. Thorax. 2021 Jan;76(1):61-63. doi: 10.1136/thoraxjnl-2020-215042. Epub 2020 Sep 22. PMID 32963115
- [Background] Costa R, Bueno F, Albert E, Torres I, Carbonell-Sahuquillo S, Barres-Fernandez A, Sanchez D, Padron C, Colomina J, Lazaro Carreno MI, Breton-Martinez JR, Martinez-Costa C, Navarro D. Upper respiratory tract SARS-CoV-2 RNA loads in symptomatic and asymptomatic children and adults. Clin Microbiol Infect. 2021 Dec;27(12):1858.e1-1858.e7. doi: 10.1016/j.cmi.2021.08.001. Epub 2021 Aug 9. PMID 34384874
- [Background] Valle C, Martin B, Touret F, Shannon A, Canard B, Guillemot JC, Coutard B, Decroly E. Drugs against SARS-CoV-2: What do we know about their mode of action? Rev Med Virol. 2020 Nov;30(6):1-10. doi: 10.1002/rmv.2143. Epub 2020 Aug 11. PMID 32779326